CLINICAL TRIAL: NCT05243992
Title: Clinical Testing Study in Peripheral Arterial Disease (CTS-PAD)
Brief Title: Clinical Testing Study in Peripheral Arterial Disease
Acronym: CTS-PAD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Perfusio Corp. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: CTS-PAD 0133633 Ver00004.5
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Arterial Disease
Keywords: tissue perfusion; tissue hypoxemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CTS-PAD device imaging — Participants in the CTS-PAD Study will undergo a conventional ABI (cABI) evaluation, followed by the non-contact imaging evaluation with the CTS-PAD device. The supplemental CTS-PAD testing will add approximately ten (10) minutes to the overall evaluation time.

SUMMARY:
The Purpose of the Clinical Testing Study in Peripheral Arterial Disease (CTS-PAD) study is to compare measurement outcomes between conventional Ankle-Brachial Index test for Peripheral Arterial Disease with a new imaging technology from which the same data can be derived, in a series of patients referred to Vascular Surgery Clinics at the University of Rochester for suspected peripheral arterial disease.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a subset of peripheral vascular disease, which describes a spectrum of perfusion- and metabolism-related threats to the tissues of the lower extremities. PAD affects an estimated 8.5 million adults in the US and > 200 million adults worldwide. PAD is atherosclerosis in the lower limbs, and classically results in inadequate oxygen supply to lower extremity musculature during walking. However, PAD is often asymptomatic, or symptoms are atypical. Risk factors are similar to cardiovascular and cerebrovascular diseases: smoking, diabetes, older age, high blood pressure, and high cholesterol.

The initial diagnostic evaluation step in symptomatic patients (i.e., classic claudication) with PAD is the conventional Ankle-Brachial Index (cABI) test. In symptomatic patients, an ABI < 0.90 (normal range 0.91-1.3) is approximately 72% sensitive and 99% specific for angiographically significant (> 50% stenosis) PAD. However, co-morbid diseases and asymptomatic/atypical patient characteristics adversely impact this test performance. In diabetics, this sensitivity falls to < 50%. Therefore, adequate strategies for screening asymptomatic/atypical patients presenting for PAD evaluation is an unmet healthcare need.

This Small Business Technology Transfer (STTR) Phase II observational study (CTS-PAD) objective is to test a novel technologic solution to address this need. Since cABI is a single factor test (< 0.9 = > 50% stenosis), it must be broadened to collect additional data that will increase the test specificity in this PAD sub-population. In parallel to stable ischemic heart disease and the importance of functional stenoses and myocardial microperfusion, these additional data should address end-organ tissue physiology as perfused by the atherosclerotic arterial supply. The asymptomatic patients' co-morbidities affect the tissue microvascularity (i.e., diabetes), and oxygen delivery and perfusion (i.e., smoking).

Perfusio Corp.'s Multi-spectral Physiologic Visualization (MSPV) imaging technology, now FDA-approved, is the base platform for this new approach, which in addition to dynamic perfusion analytics incorporates peripheral oxygen saturation (SpO2) and cardiovascular Vital Signs of Heart Rate (HR) and Blood Pressure (BP), all in immediate real-time. This CTS-PAD observational study device is non-invasive and non-contact.

The Hypothesis of the study is that ABI-type blood pressure ratio data and these tissue- and perfusion-related factors can be captured and integrated in real-time, to improve the sensitivity of evaluation in this PAD subset. The Objective of the CTS-PAD study is to document clinical Proof of Concept for this novel approach and device.

The CTS-PAD study is designed to simply collect these data for off-line, post-hoc analyses. The data from the CTS-PAD device will not be used for any clinical decision-making, and as such the clinical team will be blinded from the CTS-PAD device results data.

ELIGIBILITY:
Inclusion Criteria:

* patients who meet the clinical, symptomatic and or the disease complexity criteria for cABI testing
* age > 21 years
* intact bilateral upper and lower extremities

Exclusion Criteria:

* patients who are not considered candidates for the cABI test
* patients < 21 years
* women who might be pregnant or who are pregnant
* patients who are not considered eligible by the Attending Vascular Surgical team in clinic for medical reasons
* patients who are unable to undergo the cABI study
* patients who are unable to complete the precedent cABI study
* patients without intact bilateral upper and lower extremities
* patients with lower extremity edema or associated vascular disease where performance of the precedent cABI test would be difficult or unlikely to yield reliable data
* asymptomatic patients without complex disease characteristics, since they would not be referred for cABI testing

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population: The screening population for this study will be adults seen in vascular clinic referred for peripheral arterial disease. The U of R Vascular Clinic performs > 40-50 cABI studies / month, and their clinic population has patients with severe PVD at presentation, extensive cardiovascular risk factors that affect the sensitivity of cABI testing, and heterogenous age, race and gender characteristics.
  An analysis of the patient population demographics suggests that the gender distribution will be 60% male and 40% female in this study. Gender-based enrollment restrictions include women who are pregnant or who might be pregnant, since the imaging technology has not been tested in this sub-population.
  There are no enrollment restrictions based on race and/or ethnic origin. Overall enrollment is anticipated to be 60% Caucasian, 20% African-American, 6% Hispanic, non-white, 1% Asian, and 1% Other.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Ratio Comparison | ten (10) minutes
  Comparison of the cABI systolic BP threshold ratio vs. the CTS-PAD perfusion ratio

SECONDARY OUTCOMES:
Clinical status impact on CTS-PAD outcomes | ten (10) minutes
  correlate clinical status with CTS-PAD perfusion and physiologic data (SpO2, VS data)
Device use and performance | ten (10) minutes
  Evaluate device performance and patient and provider acceptance of this approach

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Ferguson, MD, Study Director — Perfusio Corp.

IPD SHARING:
Plan to Share IPD: No
All data are coded, and all analyses will be from aggregate data in the study de-identified database.

REFERENCES:
- See also: Sponsor Web site — http://www.perfusio.com